CLINICAL TRIAL: NCT06893419
Title: Definition and Testing of a New Model of Clinical Governance Based on the Integration of Tools Such as Health Technology Assessment, Clinical Practice Guidelines, Clinical Pathways, and Healthcare Performance Measurement for Planning, Implementation and Management of Healthcare Interventions in Different Settings - INTEGRATE-HEALTH-GOV - Geriatric Telemanagement of HEALTH Conditions in Nursing Home Residents Recently Discharged From the Hospital GET HEALTH-I
Brief Title: Geriatric Telemanagement of HEALTH Conditions in Nursing Home Residents Recently Discharged From the Hospital- GET HEALTH-I
Acronym: GET-HEALTH-I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INRCA_001_2025
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-03

CONDITIONS: Older Hospitalized Patients
Keywords: older patients; comprehensive geriatric assessment; nursing home; health technology assessment; telemanagement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing home residents (Experimental): A geriatric comprehensive assessment (CGA) will be conducted in nursing home residents using the data collection form by a multidisciplinary team led by the geriatrician, together with the family physician and the nursing home staff. The geriatrician will review the diagnoses, treatments, and results of the CGA. The patient will be interviewed and examined by the team, and then a multidisciplinary conference will be organized.
  Interventions: Other: Geriatric telemanagement

INTERVENTIONS:
Other: Geriatric telemanagement — The geriatrician will coordinate, through a telemedicine consultation, a team consisting of the general practitioner and the nursing home staff. The geriatrician will review the diagnoses, treatments, and results of the comprehensive geriatric assessment performed by the nursing home staff. Subsequently, the entire team will conduct a multidisciplinary conference.

SUMMARY:
Get-HEALTH-I study is a retrospective prospective interventional study to evaluate the impact of a geriatric telemanagement program on cost-effectiveness and clinical outcomes in nursing home residents post-hospital discharge.

DETAILED DESCRIPTION:
The GET HEALTH-I is a before and after study, consisting of both a retrospective and prospective component. The retrospective component of the study includes nursing home residents in the Marche region (Italy) who are readmitted to the nursing home after a hospital discharge, before the implementation of geriatric telemanagement. The prospective component, includes nursing home residents who are readmitted to the nursing home after a hospital discharge and are managed with the geriatric telemedicine intervention in addition to usual care. The primary objective of the study is to develop a geriatric co-management governance model using telemedicine for elderly patients with multimorbidity discharged from the hospital to nursing homes.The model will integrate geriatric specialists with nursing home staff and general practitioners.

A secondary objective of the study is to measure the performance of the model in terms of effectiveness and cost-effectiveness. In particular, an evaluation will be conducted on the effects of implementing the geriatric telemanagement governance model on the risk of hospitalization, geriatric syndromes (falls, delirium, pressure ulcers), number of medications, and inappropriate prescriptions. Adherence to the intervention by GPs and nursing home staff, satisfaction and perception of utility, costs, healthcare resource utilization, and cost-effectiveness will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Nursing home residents discharged from the hospital within one week of admission to the nursing home

Exclusion Criteria:

* Residents admitted for a short-term stay

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
reduction in hospitalization rate | After 6 months from baseline
  A minimum 15% reduction in the hospitalization rate will define the efficacy of the geriatric telemedicine consultation intervention

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cherubini, MD, Principal Investigator — IRCCS INRCA, Ancona, Italy
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No